CLINICAL TRIAL: NCT06449638
Title: A Multicenter, Prospective, Randomized Controlled Modified Platform Trial Assessing the Efficacy of Multiple Human Placental-Based Skin Substitutes and Standard of Care Versus SOC Alone in the Treatment of Hard-to-Heal Diabetic Foot Ulcers
Brief Title: Modified Platform Trial Assessing Multiple CAMPs and SOC Vs SOC Alone in the Treatment of Hard-to-Heal DFUs
Acronym: CAMPSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: StimLabs (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPM2401.001-M (07/24)
Record Dates: First submitted 2024-05-28; First posted 2024-06-10 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Foot Ulcer (DFU); Ulcer Foot; Diabetic Foot; Foot Ulcer
Keywords: Cellular, Acellular, Matrix-like Product (CAMP); Cellular and/or Tissue Product (CTP); Dehydrated Complete Human Placental Membrane (dCHPM)
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: CAMPSTIM employs a novel modified platform clinical trial design. CAMPSTIM will evaluate several CAMPs, specifically (4) placental-based CAMPs and Standard of Care (SOC) versus SOC alone in the treatment of nonhealing diabetic foot ulcers. The initial plan is to evaluate the four CAMPs identified in this protocol; however, the platform design allows for the inclusion of additional products which will be added following an interval analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Standard of Care (Active Comparator): Standard of care will be cleaning, debridement, ulcer moisture balance, and offloading.
  Interventions: Other: Standard of Care
- Revita (Experimental): Revita is an opaque, lyophilized dehydrated complete human placental membrane (dCHPM) allograft.
  Interventions: Other: Revita
- Relese (Experimental): Relese is a fenestrated dehydrated complete human placental membrane (dCHPM) allograft.
  Interventions: Other: Relese
- Cogenex (Experimental): Cognenex is a fenestrated dehydrated complete human placental membrane (dCHPM) allograft.
  Interventions: Other: Cogenex
- Enverse (Experimental): Enverse is a translucent dehydrated complete human placental membrane (dCHPM) allograft.
  Interventions: Other: Enverse

INTERVENTIONS:
Other: Standard of Care — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Standard of Care
Other: Revita — Participants will receive weekly applications of Revita and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Revita
Other: Relese — Participants will receive weekly applications of Relese and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Relese
Other: Cogenex — Participants will receive weekly applications of Cogenex and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Cogenex
Other: Enverse — Participants will receive weekly applications of Enverse and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Enverse

SUMMARY:
The purpose of this study is to evaluate the efficacy of four dehydrated complete human placental membrane, also defined as Cellular, Acellular, Matrix-like Products/skin substitutes, plus SOC versus SOC alone in achieving complete closure of hard-to-heal diabetic foot ulcers over 12 weeks using a modified platform trial design.

DETAILED DESCRIPTION:
The CAMPSTIM trial is a prospective, multicenter, randomized, controlled clinical trial to evaluate four separate CAMPs (Cellular, Acellular, Matrix-like Products), Revita®, Relese®, Cogenex®, and Enverse®. The study utilizes a unique modified platform trial to evaluate multiple cellular and/or tissue-based products (CTPs) in a single trial.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older.
2. Diagnosis of type 1 or 2 Diabetes mellitus.
3. At enrollment, target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 25.0 cm2 measured post debridement with the MolecuLight® Imaging Device.
4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care, prior to the initial screening visit.
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be full thickness without exposed bone.
7. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. Ankle-Brachial Index (ABI) between 0.7 and ≤ 1.3;
   2. Toe-Brachial Index (TBI) ≥ 0.6;
   3. Transcutaneous Oxygen Measurement (TCOM) ≥ 40 mmHg;
   4. Pulse Volume Resistance (PVR): biphasic.
8. If the potential subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. Target ulcers located on the plantar aspect of the foot must be offloaded for at least 14 days prior to enrollment.
10. The potential subject must consent to using the prescribed offloading method for the duration of the study.
11. The potential subject must agree to attend the weekly study visits required by the protocol.
12. The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. The potential subject is known to have a life expectancy of < 6 months.
2. The potential subject's target ulcer is not secondary to diabetes.
3. The target ulcer is infected or there is cellulitis in the surrounding skin.
4. The target ulcer exposes tendon or bone.
5. There is evidence of osteomyelitis complicating the target ulcer.
6. There is an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
7. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
8. The potential subject is taking hydroxyurea.
9. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
10. The potential subject with a previous partial amputation on the affected foot that results in a deformity that impedes proper offloading of the target ulcer.
11. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
12. The surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). MolecuLight Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
13. The surface area measurement of the Target ulcer decreases by 20% or more during the 2-week screening phase: the 2 weeks from the initial screening visit (S1) to the TV-1 visit during which time the potential subject received SOC.
14. The potential subject has an acute Charcot foot, or an inactive Charcot foot, which impedes proper offloading of the target ulcer.
15. Women who are pregnant or considering becoming pregnant within the next 6 months are excluded.
16. The potential subject has end stage renal disease requiring dialysis.
17. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.
18. A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
19. The target ulcer was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
20. The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutrition Assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The percentage of target ulcers achieving complete wound closure | 1-12 weeks
  Determine the percent of target ulcers achieving complete wound closure at 12 weeks. In addition, a qualified third-party clinician will independently confirm wound closure.

SECONDARY OUTCOMES:
Time to closure for the target ulcer | 1-12 weeks
  Time to closure will be determined for each treatment group and compared to SOC.
Percent area reduction | 1-12 weeks
  Percent Area Reduction (PAR) will be calculated from Treatment Visit (TV)-1 to Treatment Visit (TV)-13.
Adverse events | 1-14 weeks
  Incidence of adverse events will be evaluated weekly from TV-1 to the healing confirmation visit (HCV).
Change in pain in target ulcer | 1-14 weeks
  Change in target ulcer pain assessed using the Pain, Enjoyment of Life and General Activity (PEG) scale (0 to 10 where higher score indicates more severe pain and pain-related interference with life and activities) at TV-1, TV-4, TV-7, TV-10, and TV-13.
Determine improvement in Quality of Life - wQOL | 12 weeks
  Quality of Life assessed using the Wound Quality of Life (wQOL) checklist at TV-1, TV- 4, TV-7, TV- 10, and TV-13.
Determine improvement in Quality of Life - FWS | 12 weeks
  Quality of Life assessed using the Forgotten Wound Score (FWS) at TV-1, TV- 4, TV-7, TV- 10, and TV-13.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - SerenaGroup Omaha Research Center, Omaha, Nebraska
  - Wound Care of Tulsa, Tulsa, Oklahoma
  - SerenaGroup Research South, Jefferson Hills, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - SerenaGroup Monroeville, Monroeville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No